CLINICAL TRIAL: NCT02818348
Title: Clinical Trial to Evaluate Drug-drug Interactions Between Darunavir/Cobicistat and Etravirine in Hiv- Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRV/c-ETR
Record Dates: First submitted 2016-06-20; First posted 2016-06-29 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: HIV-1 Infection
Keywords: HIV infection; Darunavir/cobicistat; Etravirine, drug-drug interactions; Population PK analysis
MeSH Terms: conditions — HIV Infections | interventions — cobicistat mixture with darunavir; etravirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRV cohort (Experimental): Darunavir/Cobicistat 800/150 mg, once daily during 35 days + etravirine 400 mg, once daily during 14 days
  Interventions: Drug: darunavir/cobicistat; Drug: etravirine
- ETR cohort (Experimental): Etravirine 400 mg, once daily during 28 days + darunavir/cobicistat 800/150 mg, once daily during 7 days
  Interventions: Drug: darunavir/cobicistat; Drug: etravirine

INTERVENTIONS:
Drug: darunavir/cobicistat — 800/150 mg, once daily during 35 days + etravirine 400 mg, once daily during 14 days
  Other Names: Rezolsta
Drug: etravirine — 400 mg, once daily during 28 days + darunavir/cobicistat 800/150 mg, once daily during 7 days
  Other Names: Intelence

SUMMARY:
This study aims to provide information about the safety and pharmacokinetic drug-drug interactions between darunavir/cobicistat (800/150mg QD) and etravirine (400mg QD) in HIV-infected patients, as well as evaluate the efficacy of concomitant administration of darunavir/cobicistat and etravirine.

DETAILED DESCRIPTION:
Toxicity associated with use of nucleoside reverse transcriptase inhibitors (NRTIs) for the treatment of VIH-infection has prompted increasing interest in new antiretroviral treatment strategies without NRTIs (nuc-sparing regimens).

Ritonavir boosted protease inhibitors (PI/r) like, lopinavir, atazanavir, saquinavir and darunavir may be candidates for maintenance mono-therapy due to their high potency and genetic barrier for drug resistance and possibility for once daily dosing. However, although several controlled and uncontrolled studies have been conducted to examine the safety and tolerance of PI/r monotherapy for maintenance in HIV-infected patients, many of these studies were small or did not use controls; and evidence on the efficacy and safety of PI/r monotherapy is therefore limited. Moreover, several trials have reported a higher rate of intermittent viremia in patients with PI/r monotherapy. A metaanalysis including 10 randomised controlled clinical trials reported an absolute increase in the risk of virological failure at one year with PI/r monotherapy of roughly 10% to 13%. Therefore, PI/r monotherapy is not an option for clinicians and patients who do not want to accept such a risk.

If a nuc-sparing regimen is to be used, dual regimens may be an alternative to PI/r monotherapy. This approach could be able to prevent NRTI-derived toxicity while maintaining antiviral efficacy. Consequently, a growing interest in this strategy has emerged during recent years.

Ideally, a dual antiretroviral regimen should be efficacious and safe, it should permit once-daily administration with a low pill burden, and it should have a high genetic barrier towards the development of drug resistance mutations in patients who might eventually develop virological failure. The combination of the boosted PI darunavir plus the non-nucleoside reverse transcriptase inhibitor etravirine fulfills most of these requirements, and it may be an attractive dual antiretroviral treatment regimen. Although clinical experience with this combination is still limited, promising results from previous studies support current interest on the use of this dual therapy in clinical practice. Moreover, a fixed-dose combination (FDC) tablet containing darunavir and the new pharmacokinetic enhancer cobicistat (Rezolsta®) has been recently launched on the market. Among potential advantages, this FDC may contribute to decrease pill burden as well as to avoid medication errors. However, according to prescribing information, darunavir/cobicistat and etravirine should not be combined due to potential drug-drug interactions.

Darunavir and cobicistat are both metabolized by the isoenzyme CYP3A4 of the cytochrome P450, which is inhibited by cobicistat. On the other hand, etravirine, which is mainly metabolized by 2C19 (but also by CYP3A4 in a minor extent), is a CYP3A4 inducer. Based on this rationale, etravirine could decrease the exposure to cobicistat, eventually leading to concentrations of cobicistat which might be insufficient to boost darunavir.

Although no clinically relevant changes in drug concentrations were evidenced in specific trials evaluating the presence of drug-drug interactions between darunavir/ritonavir and etravirine, the combination of darunavir/cobicistat with etravirine might be more sensitive to the CYP3A inducing effect of etravirine. However, specific data on this potential drug-drug interaction are still lacking. Consequently, the combination of darunavir/cobicistat with etravirine is currently not recommended per prescribing until formal pharmacokinetic data supporting this combination are generated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Documented HIV infection (western blot)
3. Stable antiretroviral treatment including darunavir/cobicistat 800/150mg QD (cohort DRV) or etravirine 400mg QD (cohort ETR) for at least 4 weeks. Plasma HIV-1 RNA load <50 copies/mL for at least 12 weeks
4. In women of childbearing age*, commitment to use at least one of these birth control methods: male or female condom with or without spermicide, cap, diaphragm or sponge with or without spermicide, intrauterine device, bilateral tubal occlusion, vasectomised partner, sexual abstinence during the study.
5. Signed Informed Consent

   * According to recommendations of Clinical Trial Facilitation Group (CTFG), a woman is considered of childbearing potential: fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion Criteria:

1. Inadequate adherence to antiretroviral treatment (<90% during the last week)
2. Patients who are taking or have been taking any other medication within the last two weeks prior to be recruited in the study, including herbal medicines and food supplements, with known interactions with darunavir, cobicistat or etravirine (i.e St. John's wort, grapefruit juice, some antibiotics such as erythromycin or rifampicin; antiepileptics such as phenytoin, phenobarbital or carbamazepine; antifungals such as itraconazole or ketoconazole; antiretrovirals such as ritonavir, efavirenz or nevirapine, among others.)
3. Acute illness that could interfere with darunavir, cobicistat or etravirine pharmacokinetics (acute hepatitis…) within the prior 4 weeks
4. Active AIDS-defining illness within the prior 4 weeks
5. In women, pregnancy or breastfeeding.
6. Evidence or clinical suspicion that the patient will not be able to complete the study treatment and protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-11-23 (Actual)

PRIMARY OUTCOMES:
Darunavir, cobicistat and etravirine concentrations in plasma | on day 7 (PK1)
Darunavir, cobicistat and etravirine concentrations in plasma | on day 14 (PK2)
Darunavir, cobicistat and etravirine concentrations in plasma | on day 21 (PK2)
Grade ≥3 adverse events and serious adverse events | From baseline to 28 days follow-up (ETR cohort)
Grade ≥3 adverse events and serious adverse events | From baseline to 35 days follow-up (DRV/c cohort)

SECONDARY OUTCOMES:
HIV-1 RNA load in plasma | baseline
HIV-1 RNA load in plasma | on day 28 (ETR cohort)
HIV-1 RNA load in plasma | on day 35 (DRV/c cohort)

CONTACTS AND LOCATIONS:
Locations (1):
- Fundació Lluita contra la SIDA, Badalona, Barcelona, Spain